CLINICAL TRIAL: NCT03171467
Title: Salpingectomy in Women Undergoing Elective Laparoscopic Cholecystectomy (SaLCHE): A Feasibility Study
Brief Title: Salpingectomy at the Time of Elective Laparoscopic Cholecystectomy (SaLCHE)
Acronym: SaLCHE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Graz (Other)
Collaborators: Krankenhaus der Barmherzigen Brüder Graz (Unknown); Krankenhaus der Elisabethinen Graz (Unknown); Landeskrankenhaus Feldbach (Other); LKH Hartberg (Unknown); Krankenhaus der Barmherzigen Brüder St. Veit/Glan (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: SaLCHE
Record Dates: First submitted 2017-04-28; First posted 2017-05-31 (Actual); Last update posted 2018-04-17 (Actual); Status verified 2018-04

CONDITIONS: Prophylactic Salpingectomy; Opportunistic Salpingectomy; Laparoscopic Cholecystectomy
MeSH Terms: interventions — Salpingectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Salpingectomy (Experimental): Opportunistic salpingectomy at the time of laparoscopic cholecystectomy
  Interventions: Procedure: Salpingectomy

INTERVENTIONS:
Procedure: Salpingectomy

SUMMARY:
Prophylactic salpingectomy (also called opportunistic, risk-reducing or incidental salpingectomy) has been advocated at the time of gynecologic surgery to reduce the risk of serous ovarian cancer. This study explores the acceptability and feasibility of opportunistic salpingectomy at the time of elective laparoscopic cholecystectomy (LCHE).

DETAILED DESCRIPTION:
Many serous ovarian cancers are now thought to originate in the fimbria of the fallopian tubes. This has led a number of professional societies worldwide to recommend consideration of prophylactic salpingectomy at the time of elective gynecologic surgery or tubal sterilization.

This study explores the acceptability and feasibility of incidental (opportunistic, risk-reducing, prophylactic) salpingectomy at the time of a common nongynecologic procedure in women, i.e. elective laparoscopic cholecystectomy (LCHE). The study addresses whether women ≥45 years would accept opportunistic salpingectomy and the technical feasibility (time, port placement, complications) in women who consented to salpingectomy.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled (elective) laparoscopic cholecystectomy for a benign indication
* Age >45 years
* Consent

Exclusion Criteria:

* Age <45 years
* Desire to preserve fertility
* Cholecystectomy for malignant disease
* Extensive previous abdominal surgery

Ages: 45 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2016-08-01 (Actual); Primary Completion 2018-04-01 (Actual); Study Completion 2018-04-01 (Actual)

PRIMARY OUTCOMES:
Feasibility of opportunistic bilateral salpingectomy at the time of laparoscopic cholecystectomy | At time of laparoscopic cholecystectomy surgery
  Evaluation of how often opportunistic bilateral salpingectomy can be accomplished at the time of laparoscopic cholecystectomy

SECONDARY OUTCOMES:
Time | At the time of surgery
  Time (in minutes) from completion of cholecystectomy to completion of bilateral salpingectomy
Port repositioning | At surgery
  Rate of port repositioning
Complications | 30 days
  Number of complications due to salpingectomy
Patient-recorded outcome | Preop. and 1 year
  Bliem Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Karl F Tamussino, MD, Study Chair — Medical University of Graz
Locations (6):
- Austria (6):
  - Landeskrankenhaus Feldbach, Feldbach
  - Krankenhaus der Barmherzigen Brüder Graz, Graz
  - Krankenhaus der Elisabethinen Graz, Graz
  - Medical University of Graz, Graz
  - Landeskrankenhaus Hartberg, Hartberg
  - Krankenhaus der Barmherzigen Brüder St. Veit/Glan, Saint Veit/Glan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Long Roche KC, Abu-Rustum NR, Nourmoussavi M, Zivanovic O. Risk-reducing salpingectomy: Let us be opportunistic. Cancer. 2017 May 15;123(10):1714-1720. doi: 10.1002/cncr.30528. Epub 2017 Mar 23. PMID 28334425
- [Background] Committee opinion no. 620: Salpingectomy for ovarian cancer prevention. Obstet Gynecol. 2015 Jan;125(1):279-281. doi: 10.1097/01.AOG.0000459871.88564.09. PMID 25560145
- [Background] Falconer H, Yin L, Gronberg H, Altman D. Ovarian cancer risk after salpingectomy: a nationwide population-based study. J Natl Cancer Inst. 2015 Jan 27;107(2):dju410. doi: 10.1093/jnci/dju410. Print 2015 Feb. PMID 25628372
- [Background] Kurman RJ, Shih IeM. The Dualistic Model of Ovarian Carcinogenesis: Revisited, Revised, and Expanded. Am J Pathol. 2016 Apr;186(4):733-47. doi: 10.1016/j.ajpath.2015.11.011. PMID 27012190